CLINICAL TRIAL: NCT04926688
Title: Outcome of High-risk Breast Lesions Diagnosed on Image-guided Core Needle Biopsy: Results From a Multicenter Retrospective Study
Brief Title: High-risk Breast Lesions: A Multicenter Retrospective Study
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Aysenur Oktay, Professor, Ege University
Other Study IDs: 20-6T/41
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Premalignant Lesion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this multicenter study, the goal was to document the excisional biopsy or follow-up results of high risk lesions diagnosed on image guided CNB/VAB, and evaluate the clinical, imaging and histologic features for associated malignancy risk. The possibility of upgrade related to histologic subtype, tissue sampling and other variables was also evaluated.

DETAILED DESCRIPTION:
This is a retrospective multicentric study that include 1345 patients from 30 centers.

Patients who had a diagnosis of high risk lesions (HRL) on image guided core biopsy (tru-cut/vacuum biopsy) were reviewed in a 12 year period (between 2008 and 2020). The lesions included were ADH, LN (ALH/LCIS), papilloma (without or with atypia), RS, and FEA.

The patients who managed with an excisional biopsy or having at least 1 year follow-up documentation following the diagnosis of borderline lesion were included in the study.

Radiological findings, diameter of lesion (>15 vs <15 mm), needle biopsy type (14-16G vs 9-12G), sampling method and number of samplings (4 and >4 vs <4) were documented.

IBM SPSS Version 25.0 statistical package program was used for analysis.

ELIGIBILITY:
Study Population:

The women with diagnosis of atypical ductal hyperplasia, lobular neoplasia, flat epithelial atypia, papilloma and radial scar on image guided core needle biopsy were studied

Sampling Method: Non-Probability Sample Minimum Age: 12 Maximum Age: 86 Sex: Female Gender Based: No Accepts Healthy Volunteers: No

Criteria:

Inclusion Criteria:

* Image guided needle biopsy diagnosis
* Atypical ductal hyperplasia
* Lobular neoplasia
* Flat epithelial atypia
* Papilloma
* Radial scar
* Diagnosed on image guided needle biopsy

Exclusion Criteria:

* Fibroepithelial tumors
* Mucocele like tumors
* Diagnosed on surgical biopsy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The women with diagnosis of atypical ductal hyperplasia, lobular neoplasia, flat epithelial atypia, papilloma and radial scar on image guided core needle biopsy were studied
Sampling Method: Non-Probability Sample
Enrollment: 1345 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
upgrade rates related to histologic subtype, tissue sampling and other variables | one year
  the results from excisional biopsy or at least 1 year follow-up documentation

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Oktay, MD, Study Chair — Ege University; Ozge Aslan, MD, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After finishing statistical analysis the results will be published
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 3 months
Access Criteria: after publication